CLINICAL TRIAL: NCT00998959
Title: Feasibility and Efficacy of a Stress Reduction Intervention for Enhancing Treatment Outcome for Depressed Minority Patients
Brief Title: Stress Reduction Intervention for Enhancing Treatment Outcome for Depressed Minority Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trina E. Chang, MD (Other)
Collaborators: Dupont-Warren (Unknown)
Responsible Party: Sponsor-Investigator, Trina E. Chang, MD, Staff Psychiatrist, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008p001576
Record Dates: First submitted 2009-10-15; First posted 2009-10-21 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Major Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness based stress reduction and problem solving therapy (Experimental)
  Interventions: Behavioral: Mindfulness Based Stress Reduction and Psychoeducation
- Psychoeducation (Other)
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction and Psychoeducation — Participants will receive six individual weekly 50-minute sessions of mindfulness based stress reduction (MBSR) as well as problem solving therapy (PST. PST is a type of therapy that focuses on psychosocial problems and using your skills and resources to function better. MBSR uses exercises in mindfulness to reduce stress.
  Arms: Mindfulness based stress reduction and problem solving therapy
Behavioral: Psychoeducation — Participants will receive six individual weekly 50-minute sessions of psychoeducation. Psychoeducation consists of education on depression, its symptoms, its treatment, and recovery.
  Arms: Psychoeducation

SUMMARY:
The purpose of this study is to determine the usefulness of a stress reduction treatment in helping minority patients with major depression get better. Subjects will receive six weeks of either mindfulness-based stress reduction and problem solving therapy or psychoeducation.

DETAILED DESCRIPTION:
The purpose of this study is to determine the usefulness of a stress reduction treatment compared to psychoeducation in helping minority patients with major depression get better.

The study will last 10 weeks. During the main portion of the study, subjects will receive either individual weekly sessions of stress-reduction therapy or psychoeducation for six weeks. The stress reduction therapy will consist of mindfulness-based stress reduction and problem solving therapy, which focuses on linking psychological problems with psychosocial issues and helping you use your skills and resources to improve your functioning. The psychoeducation will consist of six sessions of education on depression and the treatment and management of symptoms. Each session will last 50 minutes, and four of the visits will also include filling out questionnaires which will take approximately 15-30 minutes to complete. One month after the last session, subjects will come in for a follow-up visit with a study clinician to see how they are doing and to fill out questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for current major depressive disorder
* Men or women aged 18-75 who self-identify as a member of a racial or ethnic minority group
* Has a PCP, therapist, psychiatrist, etc aware of their depression. Or, subject agrees to seek outside mental health treatment/management

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Feasibility (rate of enrollment, attrition) | 2 years

SECONDARY OUTCOMES:
Perceived stress | Week 10
  We will assess perceived stress at week 10 of subjects' study participation, although we allow for a 12-week period for subjects to complete the study.

CONTACTS AND LOCATIONS:
Overall Officials: Trina E. Chang, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States